CLINICAL TRIAL: NCT05203666
Title: A Multicentric Retrospective Evaluation of Clinical and Radiologic Outcome of All Patients Treated With a Removable Percutaneous Interspinous Process Spacer (LobsterProject® Techlamed®) for Symptomatic Degenerative Lumbar Spinal Stenosis in 2019.
Brief Title: Clinical and Radiological Outcomes Following Insertion of a Novel Removable Percutaneous Interspinous Process Spacer: an Initial Experience.
Acronym: LOBSTER
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 21Imagerie03
Record Dates: First submitted 2021-12-27; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-12

CONDITIONS: Degenerative Lumbar Spinal Stenosis; Neurologic Intermittent Claudication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- degenerative lumbar spinal stenosis: All patients treated in 2019 with a percutaneous removable interspinous process spacer a neurologic intermittent clauditation due to a degenerative lumbar spinal stenosis.
  Interventions: Other: percutaneous removable interspinous process

INTERVENTIONS:
Other: percutaneous removable interspinous process — percutaneous removable interspinous process spacer a neurologic intermittent clauditation due to a degenerative lumbar spinal stenosis.

SUMMARY:
Purpose To evaluate clinical and radiologic outcome of a series of patients treated with a removable percutaneous interspinous process spacer (IPS) (LobsterProject® Techlamed®) for symptomatic degenerative lumbar spinal stenosis (DLSS).

Methods All patients treated in the two considered Centres with this IPS during 2019 were retrospectively reviewed. Patients with incomplete clinical or radiological documentation were not included. Procedures were performed under deep sedation or general anaesthesia by two interventional radiologists. Patients were clinically evaluated before intervention and at 3-month follow-up with Visual Analog Scale for pain (VAS), Oswestry Disability Index (ODI) and radiologically with MRI or CT scans. Neural foramina were independently measured for each patient on pre- and post-procedural CT scans by two radiologists.

ELIGIBILITY:
Inclusion Criteria:

* removable percutaneous IPS treatment
* attended interventional radiology outpatient consultations for back pain and NIC, refractory to medical treatment

Exclusion Criteria:

* PS positioning included cauda equina syndrome
* permanent motor deficit,
* previous spine surgery,
* spondylolisthesis greater than Meyerding grade I,
* local or systemic infection and severe osteoarthritis with pronounced osteophytosis or bone bridges

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated with this removable percutaneous IPS in our two Centres from December 2018 to February 2020 were retrospectively reviewed and those with complete imaging and clinical data were selected. Patients attended interventional radiology outpatient consultations for back pain and NIC, refractory to medical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | Baseline
  Disability level evaluated with Oswestry Disability Index before intervention
Oswestry Disability Index | 3 Months
  Disability level evaluated with Oswestry Disability Index after intervention

SECONDARY OUTCOMES:
Visual Analog Scale for pain | Baseline
  Pain level from 0 (no pain) to 100 (unbearable pain) before intervention
Visual Analog Scale for pain | 3 Months
  Pain level from 0 (no pain) to 100 (unbearable pain) after intervention
Variation of foraminal area | Baseline
  Variation of cross sectional area of neural foramina of the treated level on pre-procedural and post-rocedural CT scan
Variation of foraminal area | 3 Months
  Variation of cross sectional area of neural foramina of the treated level on pre-procedural and post-rocedural CT scan

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pavan LJ, Dalili D, De Vivo AE, Hamel-Senecal A, Torre F, Rudel A, Manfre L, Amoretti N. Clinical and radiological outcomes following insertion of a novel removable percutaneous interspinous process spacer: an initial experience. Neuroradiology. 2022 Sep;64(9):1887-1895. doi: 10.1007/s00234-022-02977-y. Epub 2022 May 31. PMID 35641830